CLINICAL TRIAL: NCT06424873
Title: Dynamic Whole-body PET/CT Imaging in Clinical Oncology
Acronym: Dynamic PET/CT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Valentina Garibotto (Other)
Responsible Party: Sponsor-Investigator, Valentina Garibotto, Head of the Division of Nuclear Medicine and Molecular imaging, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-02102
Record Dates: First submitted 2023-11-09; First posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Fluorodeoxyglucose F18; proto-oncogene protein c-fes-fps

STUDY DESIGN:
Intervention Model Description: PET/CT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- One arm study (Experimental): Additionnal images during PET/CT
  Interventions: Radiation: PET/CT with FDG or FES

INTERVENTIONS:
Radiation: PET/CT with FDG or FES — The study consists of an additional 50 minutes of imaging during the radiotracer's uptake phase prior to their clinical scan (standard of care).

SUMMARY:
The goal of this clinical trial is to to achieve robust quantitative whole- body parametric imaging in clinically feasible scan times in patient with oncologic pathology .

The main question[s] it aims to answer are:

* [question 1]
* [question 2] Participants will [describe the main tasks participants will be asked to do, treatments they'll be given and use bullets if it is more than 2 items].

DETAILED DESCRIPTION:
Whole body hybrid PET/CT imaging, making use of the standardized uptake value (SUV), is well established in clinical setting for diagnosis and staging, treatment response monitoring and radiation therapy treatment planning of a wide range of oncologic malignancies. However, the SUV metric derived from static PET data does not capture the dynamics of the PET probe biodistribution in the body.

The present work proposes to fill in this notable gap: namely to merge whole-body and dynamic PET/CT imaging, to achieve robust quantitative whole- body parametric imaging in clinically feasible scan times. Our proposed approach has the potential to significantly enhance diagnostic, prognostic and treatment response monitoring capabilities of PET/CT and to fundamentally alter routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Patients clinically indicated for whole-body PET evaluation.
2. Patient must agree to lie still in the camera.
3. Patient must be able to comply with study procedures.
4. Patient must be able to provide informed consent.

Exclusion Criteria:

1. Patients < 18 years of age.
2. Pregnant women are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Standard SUV measurement metric | through study completion , an average of 2 years
  The standard SUV measurement metric will be compared with the measured influx rate Ki as obtained from dynamic PET/CT imaging for FDG-avid processes. We expect a correlation coefficient of at least 0.8.

SECONDARY OUTCOMES:
Image quality | through study completion , an average of 2 years
  This will be assessed by clinical PET/CT readers, on a 5 point scale.
Certainty in diagnosis of FDG-avid processes | through study completion , an average of 2 years
  This will be assessed by clinical PET/CT readers, on a 5 point scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Geneva University Hospitals, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No